CLINICAL TRIAL: NCT03592056
Title: Incidence of Hemidiaphragmatic Paralysis Using 0.04% Levobupivacaine for Continuous Interscalene Brachial Plexus Blocks in Arthroscopic Shoulder Surgeries
Brief Title: Hemidiaphragmatic Paralysis With Diluted Continuous Interscalene Plexus Infusions
Status: Terminated | Type: Observational
Why Stopped: interim analysis proved that protocol intervention had no preventive effect
Sponsor: Clinica las Condes, Chile (Other)
Responsible Party: Principal Investigator, Julián Aliste, Anesthesiololgist, Clinical Instructor, Clinica las Condes, Chile
Other Study IDs: MA012018
Record Dates: First submitted 2018-07-06; First posted 2018-07-19 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Diaphragmatic Paralysis; Postoperative Pain; Acute Pain; Shoulder Pain; Shoulder Injury
Keywords: hemidiaphragmatic paralysis; continuous plexus block; interscalene plexus block; diluted local anesthetic infusion; ambulatory regional analgesia; ambulatory continuous nerve block; continuous local anesthetic infusion
MeSH Terms: conditions — Respiratory Paralysis; Pain, Postoperative; Acute Pain; Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interscalene brachial plexus block (ISB) constitutes the analgesic criterion standard for shoulder surgery. However, it is associated with a high incidence of hemidiaphragmatic paralysis (HDP) that may not be tolerated by patients with chronic pulmonary disease. Continuous ISBs have not avoided this complication with the reported and regularly used local anesthetic dilutions (i.e. 0.125% bupivacaine, 0.25% ropivacaine, etc). This observational study will register the incidence of HDP in continuous interscalene block (CISB) using a very diluted solution of levobupivacaine (0.04%) in patients undergoing arthroscopic shoulder surgery.

The main objective of this study is to determine the frequency of HDP the first postoperative day before patient discharge(POD).

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 35

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to local anesthetics (LAs)
* pregnancy
* prior surgery in the ipsilateral neck region
* chronic pain conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing arthroscopic shoulder surgery and programmed to receive a continuous interscalene block as part of postoperative analgesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Hemidiaphragmatic paralysis before discharge | 24 hours after surgery
  Defined as less than 25% of basal diaphragm excursion evaluated with ultrasonography

SECONDARY OUTCOMES:
Hemidiaphragmatic paralysis after surgery | 30 minutes after arrival to post anesthetic care unit (PACU)
  Defined as less than 25% of basal diaphragm excursion evaluated with ultrasonography
Amount of local anesthetic (LA) boluses used before discharge. | 24 hours after surgery
  boluses of LA administered by the patient controlled infusor in adidiotn to a basal rate.
Level of static postoperative pain at 30 minutes of arrival to PACU | 30 minutes after arrival to PACU
  level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static postoperative pain 1 hour after arrival to PACU | 60 minutes after arrival
  level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static postoperative pain 3 hour after arrival to PACU | 3 hours after arrival to PACU
  level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
level of static pain 6 hours after arrival to PACU | 6 hours after arrival to PACU
  level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static pain 12 hours after arrival to PACU | 12 hour after arrival to PACU
  Level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static pain before discharge | 24 hours post surgery
  Level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static pain during first day after the day of discharge | 48 hours after surgery
  Level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
Level of static pain during second day after the day of discharge | 72 hours after surgery
  Level of pain at rest referred by the patient using a numeric rating scale from 0 to 10
intraoperative morphine equivalent consumption | intraoperative period
  total amount of morphine equivalent opioid requirement in milligrams
postoperative morphine equivalent consumption | 24 hours after surgery
  total amount of morphine equivalent opioid requirement in milligrams
sensory block in PACU | 30 minutes after arrival to PACU
  loss of sensation to cold in lateral deltoid area
Motor block in PACU | 30 minutes after arrival to PACU
  paresia or paralysis in operated side, shoulder, arm, forearm or hand
sensory block previous to discharge | 24 hours after surgery
  loss of sensation to cold in lateral deltoid area
motor block previous to discharge | 24 hours after surgery
  paresia or paralysis in operated side shoulder, arm, forearm or hand
Incidence of side effects before discharge | 24 hours after surgery
  presence of side effects (vascular puncture, Horner syndrome, hoarseness, LA systemic toxicity, catheter dislodgement, catheter insertion site leak), related with the block.
incidence of side effects after discharge with ambulatory continuous ISB. | 24 to 72 hours after surgery
  presence of side effects (vascular puncture, Horner syndrome, hoarseness, LA systemic toxicity, catheter dislodgement, catheter insertion site leak), related with the block.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Las Condes, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Result] Choromanski DW, Patel PS, Frederick JM, Lemos SE, Chidiac EJ. The effect of continuous interscalene brachial plexus block with 0.125% bupivacaine vs 0.2% ropivacaine on pain relief, diaphragmatic motility, and ventilatory function. J Clin Anesth. 2015 Dec;27(8):619-26. doi: 10.1016/j.jclinane.2015.03.006. Epub 2015 Jul 26. PMID 26216250
- [Result] Fredrickson MJ, Price DJ. Analgesic effectiveness of ropivacaine 0.2% vs 0.4% via an ultrasound-guided C5-6 root/superior trunk perineural ambulatory catheter. Br J Anaesth. 2009 Sep;103(3):434-9. doi: 10.1093/bja/aep195. Epub 2009 Jul 16. PMID 19608563
- [Result] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304